CLINICAL TRIAL: NCT06206538
Title: A Randomized Trial to Explore the Efficacy of Stellate Ganglion Block in Patients With Parkinson's Disease
Brief Title: Efficacy of Stellate Ganglion Block in Patients With Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: People's Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KY-0103-003
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The observation group (Experimental): The study lasted 20d for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Particularly, due to dysphagia, the patients enrolled might face difficulty in eating. For patients who were able to finish intake via mouth by compensatory means, the consistency, type, and size of food bolus was arranged. For those who cannot acquire sufficient nutrition through oral intake, the nasogastric tube feeding (NGT) was provided.
  Based on the invention above, the patients in the observation group were provided with stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g)
  Interventions: Procedure: Stellate ganglion block; Behavioral: Rehabilitation therapy
- The control group (Active Comparator): The study lasted 20d for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Particularly, due to dysphagia, the patients enrolled might face difficulty in eating. For patients who were able to finish intake via mouth by compensatory means, the consistency, type, and size of food bolus was arranged. For those who cannot acquire sufficient nutrition through oral intake, the nasogastric tube feeding (NGT) was provided.
  Interventions: Behavioral: Rehabilitation therapy

INTERVENTIONS:
Procedure: Stellate ganglion block — Based on the invention above, the patients in the observation group were provided with Stellate ganglion block , using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block . The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: The observation group
Behavioral: Rehabilitation therapy — he study lasted 20d for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training and nutrition support.
  Particularly, due to dysphagia, the patients enrolled might face difficulty in eating. For patients who were able to finish intake via mouth by compensatory means, the consistency, type, and size of food bolus was arranged. For those who cannot acquire sufficient nutrition through oral intake, the nasogastric tube feeding (NGT) was provided.
  Other Names: Rehabilitation Treatment

SUMMARY:
The goal of this or clinical trial is to explore efficacy of stellate ganglion block on dysphagia and activities of daily living in patients with Parkinson's disease. The main question it aims to answer are:

• Can stellate ganglion block improve the dysphagia and activities of daily living in patients with Parkinson's disease.

Participants will be divided into the the control group and observation group evenly. All the patients were provided with routine therapy, while the patients in the observation group were given stellate ganglion block. The swallowing function, and activities of daily living of the two groups of patients before and after treatment were evaluated.

DETAILED DESCRIPTION:
Dysphagia, or swallowing difficulty, is a common symptom associated with Parkinson's disease. It is characterized by weakened chewing and throat muscles, leading to difficulties in eating, coughing, and a sensation of choking in individuals with Parkinson's disease.

The goal of this or clinical trial is to explore efficacy of stellate ganglion block on dysphagia and activities of daily living in patients with Parkinson's disease. The main question it aims to answer are:

• Can stellate ganglion block improve the dysphagia and activities of daily living in patients with Parkinson's disease.

Participants will be divided into the the control group and observation group evenly. All the patients were provided with routine therapy, while the patients in the observation group were given stellate ganglion block. The swallowing function, and activities of daily living of the two groups of patients before and after treatment were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Meeting the diagnostic criteria for Parkinson's disease developed by the Neurology Branch of the Chinese Medical Association in 2006.
* Diagnosed with dysphagia confirmed by the video fluoroscopic swallowing study.
* Stable vital signs, conscious, able to cooperate with assessment and treatment.

Exclusion Criteria:

* Dysphagia possibly caused by other reasons, such as cerebrovascular disease, trauma, neuromuscular diseases, malignant diseases of the pharynx and larynx, and digestive tract diseases.
* History of mental diseases or use of antipsychotics.
* Complicated with cognitive impairment or consciousness dysfunction.
* Simultaneously suffering from severe liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 20
  On the day 1 and day 20, Penetration-Aspiration Scale is used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food enter the airway and caused penetration or aspiration during the swallowing process. As the level increases, the severity of dysphagia also increases.The scores rang from 0 to 8

SECONDARY OUTCOMES:
Modified Barthel Index | day 1 and day 20
  On the day 1 and day 20, the activities of daily living of patients will be assessed using the modified Barthel Index . The scale includes 10 items such as feeding, bathing, walking, dressing. Each item is rated on a 4-point scale based on the level of assistance required, with a total score of 100 points. There is a positive correlation between activities of daily living and the final score.
Swallowing duration | day 1 and day 20
  The time duration that the patient swallowed the contrast agent under Videofluoroscopic Swallowing Study the is recorded.Unit: seconds.
Functional Oral Intake Scale | day 1 and day 20
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Zheng Da yi Yuan Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No